CLINICAL TRIAL: NCT06760364
Title: A Single-Arm, Open-Label, Phase I Study of CHT102 for MSLN-Positive Advanced Pancreatic Cancer
Brief Title: A Clinical Study of CHT102 in MSLN-Positive Advanced Pancreatic Cancer
Acronym: CHAMPION
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Nanjing Calmhome Cell and Gene Engineering Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT102SIIT-02
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-11

CONDITIONS: Advanced Pancreatic Cancers
Keywords: Allogeneic CAR-T; Safety; Efficacy; PK

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHT102 infusion (Experimental): CHT102 will be dosing by arterial infusion.
  Interventions: Drug: CHT102

INTERVENTIONS:
Drug: CHT102 — CHT 102 : MSLN UCAR-T.

SUMMARY:
Evaluate the safety and efficacy of mesothelin-targeting UCAR-T cells in the treatment of mesothelin-positive advanced pancreatic cancer

DETAILED DESCRIPTION:
3 planned dose cohorts will be evaluated during dose escalation phase. The dose expansion will be initiated after SRC (safety review committee) review the avaliable safety, PK and preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign a written informed consent documen；
2. At the date of signing ICF, 18 ~70 years old, male or female；
3. Histopathological confirmed advanced or metastatic pancreatic cancer patients who have failed to standard treatment or intolerance with standard treatment；
4. Positive mesothelin expression;
5. At least one measurable lesion at baseline per RECIST version 1.1；
6. The expected survival time is more than 12 weeks;
7. ECOG 0-1 points;
8. Adequate organ functions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2027-12-24 (Estimated); Study Completion 2039-12-24 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years
  Treatment-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 4 weeks, and overall
  The total response rate after 90 days of treatment with study drug.
Disease control rate (DCR) | At 4 weeks, and overall
  The disease control rate after 90 days of treatment with study drug.
Progress-free survival(PFS) | 2 years
  PFS will be assessed from the first CHT102 infusion to death from any cause or the first assessment of progression (Assessed based on RECIST criteria)
Overall survival (OS ) | 3 years
  OS will be assessed from the first CHT102 infusion to death from any cause (Assessed based on RECIST criteria)
pharmacokinetics (PK) | 6 months
  Concentration levels of MSLN+ CAR-T cells
PD | 6 months
  Concentration levels of MSLN U CAR-T-related serum cytokines, such as IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α, etal

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No